CLINICAL TRIAL: NCT06852716
Title: A Study of Behavioural Change in Elderly Patients With Chronic Obstructive Pulmonary Disease on Long-term Home Oxygen Therapy Combined With Mild Cognitive Impairment Impairment: a Randomised Controlled Trial
Brief Title: A Study of in Elderly Patients With COPD on Long-term Home Oxygen Therapy Combined With MCI
Acronym: COPD、MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanjiao Yan (Other)
Responsible Party: Sponsor-Investigator, Yuanjiao Yan, Sponsor-Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LL202203
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: health education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education based on BCW theory (Experimental): It can be divided into intervention stage and follow-up stage. The intervention stage lasted for 3 months. The intervention measures in the intervention stage were as follows: stimulate the motivation to change (M), guide and motivate MCI patients to establish the health belief of insisting on long-term home oxygen therapy, and strengthen the importance and necessity of self-management; Training in behavioural change (C) Dissemination and presentation of knowledge manuals; Guide patients to correctly understand the definition, causes, clinical manifestations and hazards of COPD and MCI related diseases to improve their cognition and prevention awareness of the disease; Create a behavior change environment (O), provide a platform for patient communication, share and demonstrate home oxygen therapy skills, and improve long-term home oxygen therapy compliance. Follow-up stage: Relevant data were collected during outpatient visits or home visits to understand patients' LTHOT
  Interventions: Other: Health education based on BCW theory
- Routine health education (Active Comparator): (1) Give disease-related knowledge guidance according to nursing routine; (2) Guide patients and their families to standardize oxygen inhalation and ensure that patients correctly master oxygen inhalation operation methods; (3) Patiently answer patients' doubts about the disease, encourage patients to treat the disease with a positive attitude, and establish a good relationship of trust with patients and their families
  Interventions: Other: Routine health education

INTERVENTIONS:
Other: Health education based on BCW theory — The intervention stage lasted for 3 months. The intervention measures in the intervention stage were as follows: stimulate the motivation to change (M), guide and motivate MCI patients to establish the health belief of insisting on long-term home oxygen therapy, and strengthen the importance and necessity of self-management; Training in behavioural change (C) Dissemination and presentation of knowledge manuals; Guide patients to correctly understand the definition, causes, clinical manifestations and hazards of COPD and MCI related diseases to improve their cognition and prevention awareness of the disease; Create a behavior change environment (O), provide a platform for patient communication, share and demonstrate home oxygen therapy skills, and improve long-term home oxygen therapy compliance. Along with the Visit stage: Collect relevant data during the patient's outpatient visit or home visit to understand the patient's long-term home oxygen therapy situation.
  Arms: Health education based on BCW theory
Other: Routine health education — (1) Give disease-related knowledge guidance according to nursing routine; (2) Guide patients and their families to standardize oxygen inhalation and ensure that patients correctly master oxygen inhalation operation methods; (3) Patiently answer patients' doubts about the disease, encourage patients to treat the disease with a positive attitude, and establish a good relationship of trust with patients and their families.
  Arms: Routine health education

SUMMARY:
The goal of this clinical trial is to learn The effects of a health education programme based on BCW theory on elderly patients with chronic obstructive pulmonary disease and mild cognitive impairment The main questions it aims to answer are:Researchers will compare the effectiveness of this educational intervention with the conventional education group to see if the intervention programme can change patients' long-term home oxygen therapy adherence.The intervention phase lasts for 3 months, with sessions lasting 30 to 40 minutes, conducted twice a month. The content of both sessions is identical, resulting in a total of 6 sessions.

DETAILED DESCRIPTION:
A 2-day uniform training was conducted by the researcher herself for the other interventionists prior to the implementation of the intervention, using a combination of PPT and other A combination of PowerPoint and other written materials was used to explain the intervention process, the content of the intervention, the method of group discussion, and common problems and solutions.

The intervention process, intervention content, group discussion methods, and common problems and solutions were explained using a combination of PPT and other written materials. In order to ensure the homogeneity of the intervention, scenarios were simulated through role-playing, and the effectiveness of the training was assessed and evaluated, with problems identified and corrected.

Problems were pointed out and corrected. Elderly patients with COPD combined with MCI who met the inclusion and exclusion criteria of LTHOT were divided into 2 groups.

The patients in the experimental group received the LTHOT health education programme for elderly COPD patients with MCI based on the BCW theory, and the patients in the control group received conventional health education.

The patients in the control group received routine health education. The study subjects were divided into 2 groups, 15-20 people in each group, and the intervention activities were carried out simultaneously in the 4 groups.

The content and period of the intervention were kept consistent, and equal attention was paid to each group. 30~40min each time, 2 times a month.

The contents of the two activities are the same, a total of 6 times, the researchers carry out activities at the time agreed with the research subjects in that month, and the research subjects The researchers will carry out the activities at the agreed time with the study subjects in the same month, and the study subjects can choose the time period to participate in the health education according to their own situation.

The intervention will be carried out in the form of in-home or online health education. Group lectures will be combined with individual counselling, and individual counselling will be provided after the lectures if there are any questions.

Intervention content: Implementation of the LTHOT health education programme for elderly patients with COPD combined with MCI based on the BCW theory.

It was based on a literature review by the researchers, with reference to the Chinese Expert Consensus on Diagnosis and Treatment of Acute Exacerbation of COPD(2022 Revision) the 2022 version of the Global Strategy for the Diagnosis, Treatment and Prevention of Chronic Obstructive Lung Disease (GOLD2022 report), and so on.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years old;
* Physician-diagnosed stable COPD based on the 2022 Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines ;
* SpO₂ <88% or PaO₂ <60 mmHg;
* Met diagnostic criteria for MCI , including subjective cognitive concerns;objective cognitive impairment in memory, executive function, attention, and/or language; preserved activities of daily living ; and absence of dementia ;
* Unimpaired Mandarin communication ability ;
* Voluntary participation in the study.

Exclusion Criteria:

* comorbid asthma or malignant lung cancer;
* long-term home oxygen therapy(≥15 hours/day);
* concurrent participation in similar trials;
* significant sensory impairments, such as vision or hearing loss ; history of psychiatric disorders or congenital intellectual disabilities; comatose state, presence of major diseases, or being in the terminal stage;
* presence of other neurological diseases that could cause cognitive impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The execution of LTHOT | First and third months
  The execution of LTHOT was assessed using a self-designed Long-Term Home Oxygen Therapy Behavior Survey. Given that improper operational skills can affect the effectiveness of long-term home oxygen therapy, the survey primarily includes four dimensions: adherence to home oxygen therapy, cleaning and disinfection, safe oxygen use, and self-monitoring, with a total of 13 items. Each item has two response options: "Yes" and "No," where "Yes" indicates the behavior was performed, and "No" indicates it was not. A score of 1 is awarded for "Yes," and 0 for "No." The higher the total score, the better the patient's long-term home oxygen therapy behavior. The average daily oxygen use time was self-reported by the patient.The scores of the four dimensions were summed to obtain a total score, which was used to assess the implementation of long-term home oxygen therapy in patients.
LTHOT Health Beliefs | First and third months
  .The long-term home oxygen therapy health beliefs questionnaire designed by Yan Ying was used, with 4 dimensions and 26 items. 4 dimensions were: Perception of susceptibility to hypoxaemia，Perception of hypoxaemia severity，Perceived severity of hyepoxaemia.，Perceived benefits of long-term home oxygen therapy and Perceived barriers to long-term home oxygen therapy. According to the individual's perception of the health behavioural ability of long-term home oxygen therapy The scores were assessed according to the individual's knowledge of the health behavioural competence of long-term home oxygen therapy, with the total score ranging from 0 to 104, and the higher the score, the higher the score.

CONTACTS AND LOCATIONS:
Overall Officials: Heming Wang, Principal Investigator — Xiamen Third Hospital
Locations (1):
- Xiamen Third Hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Research data and research-related materials will be available in a repository or online. After completion of the study, relevant data will be provided in the form of a URL or DOI.
Supporting Information: SAP, Analytic Code
Time Frame: After completion of the study,relevant data will be provided in the form of a URL or DOI
Access Criteria: Researchers whose proposed use of the data has been approved

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT06852716/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT06852716/ICF_002.pdf